CLINICAL TRIAL: NCT03462121
Title: A 6-Month, Double-Blind, Phase 2 Study and 6-Month Open- Label Extension Evaluating the Safety, Tolerability, and Clinical Benefit of RPh201 in Individuals With Alzheimer's Disease With or Without Coexisting Cerebrovascular Disease
Brief Title: A Clinical Study Evaluating the Efficacy and Safety of RPh201 Treatment in Individuals With Alzheimer's Disease With or Without Coexisting Cerebrovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regenera Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-ADC-002
Record Dates: First submitted 2018-02-16; First posted 2018-03-12 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2019-06

CONDITIONS: Mild to Moderate Dementia Due to Alzheimer's Disease; With or Without Coexisting Cerebrovascular Disease
Keywords: Alzheimer's Disease,; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Cottonseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1:2
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPh201 (Experimental): A 26-week schedule consisting of twice-weekly subcutaneous administration of 400 μL of the IMP (20 mg RPh201).
  Interventions: Drug: RPh201
- Placebo (Placebo Comparator): A 26-week schedule consisting of twice-weekly subcutaneous administration of 400 μL of the vehicle control.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RPh201 — RPh201 is a well-defined extract from a botanical source
  Arms: RPh201
Other: Placebo — Inactive placebo consisting of the therapeutic vehicle
  Other Names: Cottonseed oil
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multicentre, Phase 2 study, with an optional open-label extension, to evaluate the safety, tolerability, and efficacy of RPh201 in subjects with mild to moderate AD who are eligible for enrollment in this study.

Subject participation will include a Screening Phase, Treatment Phase, and an Optional Open-Label Extension. The Screening Phase will be up to 4 weeks prior to randomization. Both the subject and their study partner(s) will sign an informed consent form (ICF). At Visit 2, Subjects will be randomized 2:1 to RPh201 or placebo. The Treatment Phase will last for 6 months post-randomization, or until subject withdrawal from the study, whichever comes first. The Optional Open-Label Extension will begin once a subject has completed the Treatment Phase and the subject and their study partner(s) have signed an ICF to continue on the study. The Optional Open-Label Extension will continue for 6 months, or until subject withdrawal from the study, whichever comes first. Subjects who do not participate in the Optional Open-Label Extension will be asked to return for an optional post-study visit 6 months after the end of the Treatment Phase.

Subjects may participate in an optional biomarker sub-study. Up to 15 subjects may also participate in an optional FDG-PET sub-study during their study participation. Separate informed consent will be required for both of these sub-studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥65 years of age at the time of consent.
* Subjects 65-69 years old, inclusive, must have evidence of cerebrovascular disease.
* Meet National Institute on Aging-Alzheimer's Association 2011 criteria for All-Cause Dementia and have evidence for probable AD or possible AD with coexisting cerebrovascular disease. Coexisting cerebrovascular disease includes evidence of any of the following: cortical infarcts, subcortical and lacunar infarcts, macro or micro-hemorrhage, and small vessel ischemic microangiopathy.
* Willing and able to provide informed consent or, if incapable of informed consent, have a legally authorized representative willing to consent on their behalf.
* MMSE at screen visit: 15-22, inclusive.
* Cholinesterase inhibitors, memantine, and other background medications impacting cognition and mood, if used, are at stable doses for at least 6 weeks prior to screening.
* A study partner is available who has adequate contact with the subject to administer study drug, oversee study drug compliance, report on adverse events (AEs), and provide meaningful input into scales and assessments.
* Adequate hearing, vision, and fluency in the language of testing.
* Magnetic resonance imaging (MRI) of the brain must reveal findings consistent with AD with or without coexisting cerebrovascular disease. In subjects for whom brain MRI is contraindicated (e.g., presence of a pacemaker), computed tomography (CT) of the brain is acceptable. Historic MRI or CT scans up to 18 months prior to screening may be used for inclusion unless there have been interval clinical events warranting an updated scan.
* Male subjects who are sexually active must agree to use one of the following acceptable methods of birth control from Screening and for at least one month after the last dose of study drug: abstinence (no sexual intercourse), male condom, or vasectomy.
* Subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Optional FDG-PET sub-study: no contraindications to PET imaging. Individuals participating in the FDG-PET sub-study will be capped at 15 volunteers and a further cap may be imposed on the number enrolling in this sub-study without evidence of cerebrovascular disease.

Exclusion Criteria:

* Neurological or non-neurological conditions other than AD and cerebrovascular disease that, in the Investigator's opinion, contribute to, or provide alternative etiology for, the subject's dementia. Examples include, but are not limited to, brain tumors, clinically significant head injury, Parkinson's disease, current or prior excess use of alcohol that, in the investigator's judgment, has caused or significantly contributed to the subject's cognitive decline, or primary psychiatric disorders (e.g., schizophrenia or bipolar affective disorder).
* Unstable medical conditions which are likely to impact subject's ability to complete the trial and which are likely to confound AE assessment. These include, but are not limited to, uncontrolled hypertension, uncontrolled diabetes, and cancer within past the 2 years. Exceptions include prostate cancer in-situ and local basal and squamous cell skin cancers.
* Chronic use of systemic or inhaled steroids (use of topical steroids is acceptable).
* Other concomitant medications that, in the Investigator's judgment, impair cognition and/or confound efficacy assessments.
* Women of child-bearing potential are excluded (e.g., women who have not been post-menopausal for at least 2 years or are not surgically sterile).
* Treatment with investigational product from a previous clinical drug trial within the last 30 days or five half-lives prior to Visit 2 (Baseline), whichever is longer.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in (Alzheimer disease assessment scale) ADAS-Cog score between Baseline and Month 6 | Month 6
  The ADAS-Cog is an established general cognitive measure scaled used in clinical trials of AD. The ADAS-Cog assesses multiple performance and cognitive domains including memory, language, praxis, and orientation. Test responses are scored using summed error points where 0 represents no errors and 70 represents errors on all items; higher scores indicate greater cognitive impairment.
Change in CDR-SB score between Baseline and Month 6 | Month 6
  The CDR is a global clinical scale with established diagnostic and severity-ranking utility widely used in clinical trials yielding global and sum of boxes scores (CDR-SB). The CDR global score is used in AD trials as a global measure of disease severity. The CDR is rated based on subject and informant input. The CDR assess three domains of cognition (memory, orientation, judgment/problem solving) and three domains of function (community affairs, home/hobbies, personal care) using semi- structured interviews of both the study subject and a companion/informant carried out by a trained rater and scored using a standard methodology. Each domain is rated on a 5-point scale of functioning as follows: (0) no impairment; (0.5) questionable impairment; (1) mild impairment; (2) moderate impairment; (3) severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). Higher scores indicate greater impairment.
AEs at Month 6 | Month 6
12-lead ECG at Month 6 | Month 6
Clinical Laboratory Assessments - (blood and urine) at at Month 6 | Month 6
  Chemistry: alkaline phosphatase, albumin, blood urea nitrogen, calcium, chloride, creatinine, glucose (random), inorganic phosphorus, potassium, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transpeptidase, lactate dehydrogenase, sodium, direct bilirubin, total bilirubin, total protein, amylase, uric acid Hematology: haemoglobin, hematocrit, red blood cell count, white blood cell (WBC) count, WBC differential (absolute counts), numerical platelet count Urinalysis: specific gravity, pH, ketones, glucose, nitrite, blood, leukocyte esterase, protein, urobilinogen, bilirubin If nitrite, blood, or protein tests are positive, a microscopic examination will be performed
Vital Signs | Month 6
  Vital signs consist of tympanic temperature, respiratory rate, blood pressure (systolic and diastolic blood pressure, mmHg), and pulse (bpm) after at least 3 minutes rest. Blood pressure will be measured in a sitting or semi-reclined seated position. Weight and height will be captured at Screening and weight will be captured at all other visits where this assessment is performed.

SECONDARY OUTCOMES:
Change from Baseline on ADAS-Cog total scores at Month 3 | Months 3
  The ADAS-Cog is an established general cognitive measure scaled used in clinical trials of AD. The ADAS-Cog assesses multiple performance and cognitive domains including memory, language, praxis, and orientation. Test responses are scored using summed error points where 0 represents no errors and 70 represents errors on all items; higher scores indicate greater cognitive impairment.
Change from Baseline on ADAS-Cog total scores at Month 5 | Month 5
  The ADAS-Cog is an established general cognitive measure scaled used in clinical trials of AD. The ADAS-Cog assesses multiple performance and cognitive domains including memory, language, praxis, and orientation. Test responses are scored using summed error points where 0 represents no errors and 70 represents errors on all items; higher scores indicate greater cognitive impairment.
Change from Baseline on ADAS-Cog total scores at Month 12 | Month 12
  The ADAS-Cog is an established general cognitive measure scaled used in clinical trials of AD. The ADAS-Cog assesses multiple performance and cognitive domains including memory, language, praxis, and orientation. Test responses are scored using summed error points where 0 represents no errors and 70 represents errors on all items; higher scores indicate greater cognitive impairment.
Change from Baseline on CDR-SB total scores at Month 3 | Month 3
  The CDR is a global clinical scale with established diagnostic and severity-ranking utility widely used in clinical trials yielding global and sum of boxes scores (CDR-SB). The CDR global score is used in AD trials as a global measure of disease severity. The CDR is rated based on subject and informant input. The CDR assess three domains of cognition (memory, orientation, judgment/problem solving) and three domains of function (community affairs, home/hobbies, personal care) using semi- structured interviews of both the study subject and a companion/informant carried out by a trained rater and scored using a standard methodology. Each domain is rated on a 5-point scale of functioning as follows: (0) no impairment; (0.5) questionable impairment; (1) mild impairment; (2) moderate impairment; (3) severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). Higher scores indicate greater impairment.
Change from Baseline on CDR-SB total scores at Month 5 | Month 5
  The CDR is a global clinical scale with established diagnostic and severity-ranking utility widely used in clinical trials yielding global and sum of boxes scores (CDR-SB). The CDR global score is used in AD trials as a global measure of disease severity. The CDR is rated based on subject and informant input. The CDR assess three domains of cognition (memory, orientation, judgment/problem solving) and three domains of function (community affairs, home/hobbies, personal care) using semi- structured interviews of both the study subject and a companion/informant carried out by a trained rater and scored using a standard methodology. Each domain is rated on a 5-point scale of functioning as follows: (0) no impairment; (0.5) questionable impairment; (1) mild impairment; (2) moderate impairment; (3) severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). Higher scores indicate greater impairment.
Change from Baseline on CDR-SB total scores at Month 12 | Month 12
  The CDR is a global clinical scale with established diagnostic and severity-ranking utility widely used in clinical trials yielding global and sum of boxes scores (CDR-SB). The CDR global score is used in AD trials as a global measure of disease severity. The CDR is rated based on subject and informant input. The CDR assess three domains of cognition (memory, orientation, judgment/problem solving) and three domains of function (community affairs, home/hobbies, personal care) using semi- structured interviews of both the study subject and a companion/informant carried out by a trained rater and scored using a standard methodology. Each domain is rated on a 5-point scale of functioning as follows: (0) no impairment; (0.5) questionable impairment; (1) mild impairment; (2) moderate impairment; (3) severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). Higher scores indicate greater impairment.
Change from Baseline in ADCS-ADL total score at Month 3 | Month 3
  The ADCS-ADL is an assessment consisting of 23 basic and instrumental ADLs used in mild to moderate AD subjects.7 The scores of the informant-rated assessment are graded against a 78- point scale, with lower scores indicating greater impairment.
Change from Baseline in ADCS-ADL total score at Months 12 | Month 12
  The ADCS-ADL is an assessment consisting of 23 basic and instrumental ADLs used in mild to moderate AD subjects.7 The scores of the informant-rated assessment are graded against a 78- point scale, with lower scores indicating greater impairment.
Change from Baseline in NPI total score at Month 3 | Month 3
  The NPI is designed to detect, quantify, and track changes of psychiatric symptoms in a demented population.6 It uses a structured, caregiver-based interview format to assess 10 behavioral domains (delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, apathy, irritability, euphoria, disinhibition, and aberrant motor behavior). The same behaviors are then rated on level of severity (1 = mild, 2 = moderate, 3 = severe). The domain total score is the product of the frequency score multiplied by the severity score for that behavioral domain. An NPI total score is obtained by summing all the individual domain total scores.
Change from Baseline in NPI total score at Month 6 | Month 6
  The NPI (Appendix 7) is designed to detect, quantify, and track changes of psychiatric symptoms in a demented population.6 It uses a structured, caregiver-based interview format to assess 10 behavioral domains (delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, apathy, irritability, euphoria, disinhibition, and aberrant motor behavior). The same behaviors are then rated on level of severity (1 = mild, 2 = moderate, 3 = severe). The domain total score is the product of the frequency score multiplied by the severity score for that behavioral domain. An NPI total score is obtained by summing all the individual domain total scores.
Change from Baseline in NPI total score at Month 12 | Month 12
  The NPI (Appendix 7) is designed to detect, quantify, and track changes of psychiatric symptoms in a demented population.6 It uses a structured, caregiver-based interview format to assess 10 behavioral domains (delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, apathy, irritability, euphoria, disinhibition, and aberrant motor behavior). The same behaviors are then rated on level of severity (1 = mild, 2 = moderate, 3 = severe). The domain total score is the product of the frequency score multiplied by the severity score for that behavioral domain. An NPI total score is obtained by summing all the individual domain total scores.
Change from Baseline in the MMSE at Month 3 | Month 3
  The MMSE is a brief 30-point examination consisting of 11 questions intended to evaluate an adult subject's level of cognition. The MMSE evaluates 6 areas of cognition: orientation, attention, immediate recall, short-term recall, language, and the ability to follow simple verbal and written commands. In addition, it provides a total score allowing the examiner to evaluate the severity of cognitive impairment.
  The MMSE will be scored using backward spelling (WORLD) and not serial subtractions. The scoring of WORLD will follow the original Folstein et al (1975)8 instructions for this assessment.
Change from Baseline in the MMSE at Month 6 | Month 6
  The MMSE is a brief 30-point examination consisting of 11 questions intended to evaluate an adult subject's level of cognition. The MMSE evaluates 6 areas of cognition: orientation, attention, immediate recall, short-term recall, language, and the ability to follow simple verbal and written commands. In addition, it provides a total score allowing the examiner to evaluate the severity of cognitive impairment.
  The MMSE will be scored using backward spelling (WORLD) and not serial subtractions. The scoring of WORLD will follow the original Folstein et al (1975)8 instructions for this assessment.
Change from Baseline in the MMSE at Month 12 | Month 12
  The MMSE is a brief 30-point examination consisting of 11 questions intended to evaluate an adult subject's level of cognition. The MMSE evaluates 6 areas of cognition: orientation, attention, immediate recall, short-term recall, language, and the ability to follow simple verbal and written commands. In addition, it provides a total score allowing the examiner to evaluate the severity of cognitive impairment.
  The MMSE will be scored using backward spelling (WORLD) and not serial subtractions. The scoring of WORLD will follow the original Folstein et al (1975)8 instructions for this assessment.
AEs at Month 12 | Month 12
Clinically significant changes in vital signs at Month 12 | Month 12
12-lead ECG at Month 12 | Month 12
Clinical Laboratory Assessments - (blood and urine) at Month 12 | Month 12
  Chemistry: alkaline phosphatase, albumin, blood urea nitrogen, calcium, chloride, creatinine, glucose (random), inorganic phosphorus, potassium, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transpeptidase, lactate dehydrogenase, sodium, direct bilirubin, total bilirubin, total protein, amylase, uric acid Hematology: haemoglobin, hematocrit, red blood cell count, white blood cell (WBC) count, WBC differential (absolute counts), numerical platelet count Urinalysis: specific gravity, pH, ketones, glucose, nitrite, blood, leukocyte esterase, protein, urobilinogen, bilirubin If nitrite, blood, or protein tests are positive, a microscopic examination will be performed
Vital Signs | Month 12
  Vital signs consist of tympanic temperature, respiratory rate, blood pressure (systolic and diastolic blood pressure, mmHg), and pulse (bpm) after at least 3 minutes rest. Blood pressure will be measured in a sitting or semi-reclined seated position. Weight and height will be captured at Screening and weight will be captured at all other visits where this assessment is performed.

OTHER OUTCOMES:
AD blood biomarkers to assess change from Baseline at Month 6 | Month 6
AD blood biomarkers to assess change from Baseline at Month 12 | Month 12
Change in FDG-PET between Baseline and Month 6 in a subset of subjects (Optinal) | Month 6
  18-Fluoro-deoxyglucose positron emission tomography (FDG-PET) is a noninvasive, 3-dimensional imaging modality that has become widely used in the management of subjects with malignant lymphomas.9 Up to 15 subjects will participate in an optional FDG-PET sub-study to assess the effect of RPh201 on cerebral glucose metabolism at Baseline and after 6 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cohen, MD, Principal Investigator — Toronto Memory Program
Locations (5):
- Canada (5):
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Gerontion Research Inc., The Center for Memory & Aging, Toronto, Ontario
  - Recherches Neuro-Hippocampe Inc. d/b/a Clinique de la Memoire de l'Outaouais, Gatineau, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided